CLINICAL TRIAL: NCT01110447
Title: Secondary Prophylaxis of Hepatic Encephalopathy: A Double Blind, Randomized, Placebo Controlled Study With Supplementation With a Probiotic Preparation
Brief Title: Secondary Prophylaxis of Hepatic Encephalopathy With a Probiotic Preparation
Acronym: VSL#3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CD Pharma India Pvt. Ltd. (Industry)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MHE2-VSL#3-Ver3_30032010
Record Dates: First submitted 2010-04-23; First posted 2010-04-26 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy, probiotics
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 (Experimental): VSL#3® is made up of 4 strains of Lactobacilli (L. paracasei, L. plantarum, L. acidophilus and L. delbrueckii subsp. bulgaricus), 3 strains of Bifidobacteria (B. longum, B. infantis, B. breve) and 1 strain of Streptococcus thermophilus.
  Interventions: Drug: VSL#3
- Placebo (Placebo Comparator): Placebo sachets contain corn starch
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VSL#3 — VSL#3® is made up of 4 strains of Lactobacilli (L. paracasei, L. plantarum, L. acidophilus and L. delbrueckii subsp. bulgaricus), 3 strains of Bifidobacteria (B. longum, B. infantis, B. breve) and 1 strain of Streptococcus thermophilus. Dose would be 1 sachet per day (Each sachet containing 900 Billion CFU). The duration of treatment would be for 24 weeks
  Other Names: Probiotic
  Arms: VSL#3
Other: Placebo — Placebo sachets contain corn starch. Dose: 1 sachet per day Duration of treatment: 24 weeks
  Other Names: Dummy Preparation
  Arms: Placebo

SUMMARY:
The aim of the proposed project is to study the effects of a probiotic preparation (VSL#3®) for the prevention of recurrence of HE (Hepatic encephalopathy) in patients after the recovery of an episode of overt HE (secondary prophylaxis)

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) represents a spectrum of neuropsychiatric abnormalities seen in patients with liver dysfunction after exclusion of other known brain disease. The Working Party at the 11th World Congress of Gastroenterology, Vienna proposed a multi-axial definition of HE that defined both, the type of hepatic abnormality (type A, B or C) and the duration/characteristics of neurological manifestations (episodic, persistent or minimal HE) in chronic liver disease. Overt hepatic encephalopathy occurs in 30%-45% of cirrhotic patients and 10%-50% of patients with transjugular intrahepatic portosystemic shunt. Development of HE is associated with a poor prognosis. Bustamante et al reported the survival probability of 42% at 1 year of follow-up and 23% at 3 years in patients with cirrhosis with a first episode of acute HE. The primary treatment of HE is the identification and treatment of the precipitating factors. The majority of the drugs used in the treatment of HE are primarily directed at the reduction or elimination of the increased neurotoxic ammonia levels. A meta-analysis of 22 randomized trials highlighted the lack of data supporting the efficacy of nonabsorbable disaccharides; however, the investigators concluded that current evidence is insufficient to support or refute the use of nonabsorbable disaccharides for treatment of HE. Recent studies with well defined groups however demonstrated the efficacy of lactulose. Alternative therapies such as benzodiazepine receptor antagonists, branched-chain amino acids, and L-ornithine-L-aspartate also have been shown to have some role. Antibiotics are effective in the treatment of HE, but adverse effects and concerns about long-term safety have limited their widespread use. Probiotics may have multiple beneficial effects in the prevention and/or treatment of HE. All four published studies on the effect of probiotics on hepatic encephalopathy have demonstrated efficacy. Treating patients to prevent development of a first episode is classified as primary prophylaxis of HE and preventing recurrence of HE in patients who had a previous episode of HE as secondary prophylaxis of HE. Sharma et al recently demonstrated that lactulose is effective in secondary prevention of HE. This study will assess the effects of a probiotic preparation for the prevention of recurrence of HE (secondary prophylaxis) in patients after the recovery of an episode of overt HE.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having cirrhosis of liver at the Inpatient/Outpatient Liver Clinic of Department of Hepatology, PGIMER, Chandigarh, will be candidates for enrollment.
* The diagnosis of cirrhosis of liver will be based on clinical, biochemical, and ultrasonographical or liver histological data.

Exclusion Criteria:

* Alcohol intake during the past 6 weeks
* Hepatocellular carcinoma
* Previous transjugular intrahepatic portosystemic shunt or shunt surgery
* Significant comorbid illness such as heart, respiratory, or renal failure
* Any neurologic diseases such as Alzheimer's disease, Parkinson's disease, and nonhepatic metabolic encephalopathies.
* Patients on psychoactive drugs, such as antidepressants or sedatives
* Those who restart alcohol consumption during follow-up will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary end point will be development of overt HE or completion of a follow-up of 6 months after enrollment | 6 months after enrollment

SECONDARY OUTCOMES:
Improvement in liver functions (Child and MELD score), psychometry (psychometric hepatic encephalopathy score), blood ammonia, blood cytokines level and survival time after medication | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Radha K Dhiman, MD,DM,MNAMS, Principal Investigator — Postgraduate Institute of Medical Education & Research (PGIMER)
Locations (1):
- Dept. of Hepatology, PGIMER, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Dhiman RK, Grover GS, Premkumar M, Roy A, Taneja S, Duseja A, Arora S; MMPHCRF Investigators. Outcomes of Real-World Integrated HCV Microelimination for People Who Inject Drugs: An expansion of the Punjab Model. EClinicalMedicine. 2021 Oct 17;41:101148. doi: 10.1016/j.eclinm.2021.101148. eCollection 2021 Nov. PMID 34712928
- [Derived] Dhiman RK, Grover GS, Premkumar M, Taneja S, Duseja A, Arora S, Rathi S, Satsangi S, Roy A; MMPHCRF Investigators. Decentralized care with generic direct-acting antivirals in the management of chronic hepatitis C in a public health care setting. J Hepatol. 2019 Dec;71(6):1076-1085. doi: 10.1016/j.jhep.2019.07.006. Epub 2019 Jul 17. PMID 31325468
- [Derived] Dhiman RK, Rana B, Agrawal S, Garg A, Chopra M, Thumburu KK, Khattri A, Malhotra S, Duseja A, Chawla YK. Probiotic VSL#3 reduces liver disease severity and hospitalization in patients with cirrhosis: a randomized, controlled trial. Gastroenterology. 2014 Dec;147(6):1327-37.e3. doi: 10.1053/j.gastro.2014.08.031. Epub 2014 Aug 27. PMID 25450083